CLINICAL TRIAL: NCT07079267
Title: Olpasiran Expanded Access Program
Status: Available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: Olpasiran Expanded Access
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

MeSH Terms: interventions — olpasiran

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Olpasiran

SUMMARY:
Expanded access requests for Olpasiran may be considered for adult participants with elevated Lp(a) and atherosclerotic cardiovascular disease (ASCVD). To request access, use Responsible Party contact information provided in this record.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years
Age Groups: Adult, Older Adult